CLINICAL TRIAL: NCT06112223
Title: Preemptive Oral Gabapentin Versus Tramadol on Postoperative Pain After Knee Arthroscopy Done Under Spinal Anesthesia: A Prospective Randomized Trial
Brief Title: Preemptive Oral Gabapentin and Tramadol on Postoperative Pain After Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Laila Elahwal, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR151/3/23
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Gabapentin; Tramadol; Postoperative Pain; Knee Arthroscopy; Spinal Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): Patients will receive oral gabapentin 600 mg 1 hour before the surgery.
  Interventions: Drug: Gabapentin
- Tramadol (Experimental): Patients will receive oral tramadol 100 mg 1 hour before the surgery.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Gabapentin — Patients will receive oral gabapentin 600 mg 1 hour before the surgery.
  Arms: Gabapentin
Drug: Tramadol — Patients will receive oral tramadol 100 mg 1 hour before the surgery.
  Arms: Tramadol

SUMMARY:
The aim of this study to evaluate the effect of preemptive oral gabapentin versus tramadol on postoperative pain after knee arthroscopy under spinal anesthesia.

DETAILED DESCRIPTION:
Orthopedic surgeries are frequently associated with moderate-to-severe postoperative pain that can decrease mobility in the immediate postoperative period, interfere with postoperative rehabilitation, and delay hospital discharge. Pain may also become chronic.

Spinal anesthesia is the most popular anesthesia technique worldwide in orthopedic lower limb surgeries. However, its relatively short duration of action may limit the excellent postoperative analgesic effect. Thus, many adjuvants had been used to improve postoperative analgesia and decrease consumption of postoperative analgesics.

Gabapentin is a gamma aminobutyric acid analogue that is known as an anticonvulsant drug. This drug is tolerated well and has known effects on pain and anxiety.

Tramadol, a commonly used postoperative analgesic, is a synthetic centrally acting opioid analgesic. The various actions include inhibition of noradrenaline and serotonin reuptake, and also inhibition of M1 and M3 muscarinic receptors

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old.
* Both sexes. American Society of Anesthesiologists (ASA) physical status I and II
* Undergoing knee arthroscopy procedures.
* under spinal anesthesia.

Exclusion Criteria:

* Cardiac patients.
* Patients with known allergy to drug of study.
* Prolonged administration of NSAIDS or other analgesics due to chronic pain of any reason.
* Cirrhosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The intensity of postoperative pain | 24 hours postoperatively
  Assessment of postoperative pain will be done with a analogue scale (VAS; 0=no pain and 10=worst possible pain). At discharge post-operative and every 2 hours postoperative till 12hours then every 6 hours for the first 24 hours.

SECONDARY OUTCOMES:
The total amount of morphine consumption in the first 24-hour postoperative | 24 hours postoperatively
  Rescue analgesia in the form of 3 mg of IV morphine will be given if the visual analog scale (VAS) score> 3.
The time first rescue analgesia | 24 hours postoperatively
  Rescue analgesia in the form of 3 mg of IV morphine will be given if the visual analog scale (VAS) score≥ 4.
The incidence of side effects | 24 hours postoperatively
  Any undesirable side effects during the first 24 hours will be recorded such as as nausea, vomiting &hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.